CLINICAL TRIAL: NCT01272921
Title: A Dose Response Study for Duration of Analgesia Using Bupivacaine and Ropivacaine for Infragluteal Parabiceps Sciatic Block
Brief Title: The Use of Bupivacaine and Ropivacaine for Sciatic Nerve Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Antoun Nader, Professor in Anesthesiology and Orthopaedic Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STU00035380
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: The Duration of Motor Block May Vary Between 12-36 Hrs
MeSH Terms: interventions — Bupivacaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Active Comparator): Varying does to determine duration of analgesia following a sciatic nerve block
  Interventions: Drug: Bupivacaine
- Ropivacaine (Active Comparator): Varying does to determine duration of analgesia following a sciatic nerve block
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Bupivacaine — Varying doses to determine the duration of analgesia
  Arms: Bupivacaine
Drug: Ropivacaine — Varying doses to determine the duration of analgesia
  Arms: Ropivacaine

SUMMARY:
The duration of motor block for infragluteal parabiceps sciatic nerve block following total knee replacement may vary between 12-36 hrs depending on the amount of local anesthetic given.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age) who are undergoing elective total knee arthroplasty will be included in the study.

Exclusion Criteria:

* Exclusion criteria for the study are patient refusal to be included in the study, contraindications to regional anesthesia, history of allergy to amide local anesthetics, the presence of a progressive neurological deficit, the presence of coagulopathy or infection, or pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoun Nader, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University, Feingberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Derived] Nader A, Kendall MC, De Oliveira GS Jr, Puri L, Tureanu L, Brodskaia A, Asher Y, Parimi V, McCarthy RJ. A dose-ranging study of 0.5% bupivacaine or ropivacaine on the success and duration of the ultrasound-guided, nerve-stimulator-assisted sciatic nerve block: a double-blind, randomized clinical trial. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):492-502. doi: 10.1097/AAP.0b013e3182a4bddf. PMID 24108248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects undergoing primary tricompartmental total knee replacement at Northwestern Memorial Hospital were asked to participate. 174 patients were approached. 142 subjects were recruited to participate.
Pre-assignment Details: Exclusion criteria: subject refusal to be included in the study, contraindications to regional anesthesia, inability to elicit an evoked motor response less than or equal to 1 mA, history of allergy to amide local anesthetics, presence of a progressive neurological deficit, opioid tolerant subjects, presence of coagulopathy, infection, or pregnancy
Groups:
- Bupivacaine: Varying does to determine duration of analgesia following a sciatic nerve block
  Bupivacaine : Varying doses to determine the duration of analgesia
- Ropivacaine: Varying does to determine duration of analgesia following a sciatic nerve block
  Ropivacaine : Varying doses to determine the duration of analgesia
Period: Overall Study
Arm/Group | Bupivacaine | Ropivacaine
Started | 71 | 71
Completed | 69 | 70
Not Completed | 2 | 1
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- GROUP 1: Varying does to determine duration of analgesia following a sciatic nerve block
  Bupivacaine : Varying doses to determine the duration of analgesia
- GROUP 2: Varying does to determine duration of analgesia following a sciatic nerve block
  Ropivacaine : Varying doses to determine the duration of analgesia
- Total: Total of all reporting groups
Arm/Group | GROUP 1 | GROUP 2 | Total
Number analyzed (Participants) | 69 | 70 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 34 | 66
  >=65 years | 37 | 36 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.93 (9.21) | 64.70 (9.26) | 65.81 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 43 | 87
  Male | 25 | 27 | 52
Region of Enrollment [Number; unit: participants]
  United States | 69 | 70 | 139

OUTCOME MEASURES:

1. Secondary Outcome: Cumulative Probabilities for Needle Positioning Above and Below CIEL.
Description: The cumulative probability distributions for the minimal current to evoke a motor response with the needle tip positioned external (above) to the common investing extraneural layer (CIEL) and the cumulative probability distribution for the needle tip postioned internal (below) to the CIEL were sought. The difference in the mean minimum threshold current (mA) for the external (above) and internal (below) CIEL positioning were calculated.
Time Frame: 1 Day
Measure: Mean (95% Confidence Interval); unit: Amplitude (mA)
Groups:
- Above CIEL: The mean threshold current required to elicit a motor response above the common investing extraneural layer (CIEL).
- Below CIEL: The mean threshold current required to elicit a motor response below the common investing extraneural layer (CIEL).
Arm/Group | Above CIEL | Below CIEL
Number analyzed (Participants) | 69 | 70
Amplitude (mA) | 0.52 [0.49 to 0.54] | 0.19 [0.18 to 0.21]
Statistical Analysis 1: Comparison: Above CIEL; Test type: Superiority or Other; p < 0.001, Z score; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [0.49 to 0.54]
Statistical Analysis 2: Comparison: Below CIEL; Test type: Superiority or Other; p < 0.001, Z score; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [0.18 to 0.21]

2. Primary Outcome: Duration of Motor and Sensory Block of the Sciatic With 0.5% Bupivacaine and Ropivacaine After Ultrasound-guided Nerve-stimulator-Assisted Needle Positioning Beneath the CIEL
Description: Subject reported and investigator measured motor and sensory blockade of the sciatic nerve with less than 10ml of 0.5% bupivacaine and ropivacaine after ultrasound-guided nerve-stimulator-assisted needle positioning beneath the common investing external layer (CIEL).
Time Frame: 3 days
Measure: Median (95% Confidence Interval); unit: Hours
Groups:
- Bupivacaine: Varying does to determine duration(motor/sensory)of analgesia following a sciatic nerve block
  Bupivacaine : 2.5ml and 5.0mL (less than 10ml) and greater than or equal to 10ml (10-30ml)
- Ropivacaine: Varying does to determine duration(motor/sensory)of analgesia following a sciatic nerve block
  Ropivacaine : 2.5ml and 5.0mL (less than 10ml) and greater than or equal to 10ml (10-30ml)
Arm/Group | Bupivacaine | Ropivacaine
Number analyzed (Participants) | 69 | 70
Hours
  Motor: < 10ml | 10 [4 to 14] | 7 [5 to 10]
  Motor: >/= 10ml | 21 [17 to 22] | 15 [14 to 15]
  Sensory: <10ml | 9 [6 to 14] | 8 [6 to 12]
  Sensory: >/= 10ml | 20 [17 to 23] | 14 [13 to 15]
Statistical Analysis 1: Comparison: Bupivacaine; The sample selected for this study,70 per drug group (or 10 in each of the 7 groups), achieves 88% power to detect a minimal difference of 4 hours in duration at a significance level (α) of 0.05 and a standard deviation of 3 hours using Williams test. We chose a difference of 4 hours as this was the interval used for assessment in the postoperative period at night. We sought to detect a difference that was equal to 1 observation period difference; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney) — Post hoc comparison were made against the 30-mL volume group and corrected for 6 comparisons using the Wilcoxon rank sum test; Mean Difference (Final Values) = -11.00, 95% CI 2-sided [-17.00 to -6.00], Standard Deviation 0
Statistical Analysis 2: Comparison: Bupivacaine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -11.00, 95% CI 2-sided [-15.00 to -6.00], Standard Deviation 0
Statistical Analysis 3: Comparison: Ropivacaine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -7.0, 95% CI 2-sided [-10.00 to -4.00], Standard Deviation 0
Statistical Analysis 4: Comparison: Ropivacaine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -6.00, 95% CI 2-sided [-7.00 to -2.00], Standard Deviation 0

ADVERSE EVENTS:
Time Frame: Time frame for adverse event reporting was 12 months following surgery.
Groups:
- GROUP 1: Varying does to determine duration(motor/sensory)of analgesia following a sciatic nerve block
  Bupivacaine : 2.5ml and 5.0mL (less than 10ml) and greater than or equal to 10ml (10-30ml)
- GROUP 2: Varying does to determine duration(motor/sensory)of analgesia following a sciatic nerve block
  Ropivacaine : 2.5ml and 5.0mL (less than 10ml) and greater than or equal to 10ml (10-30ml)
Arm/Group | GROUP 1 | GROUP 2
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/70
Other Adverse Events (participants affected / at risk) | 0/69 | 0/70

LIMITATIONS AND CAVEATS:
We used 5-mL increments of local anesthetic w/epinephrine between 5-30 mL which may have prevented from identifying more precisely the volume at which onset/duration were similar.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes